CLINICAL TRIAL: NCT06379438
Title: Treatment of Aphtous Ulcers With Photodynamic Therapy: A Randomised Controlled Clinical Trial
Brief Title: Treatment of Aphtous Ulcers With Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Cennet Neslihan Eroglu, Assoc Prof Dr, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/16022018
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Oral Ulcer; Aphthous Recurrent Ulcers
Keywords: photodynamic therapy; aphtous ulcer; indocyanine green
MeSH Terms: conditions — Oral Ulcer; Stomatitis, Aphthous | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photodynamic Therapy (PDT) Group (Experimental): Patients in the PDT group were treated in a single session on the day of admission to the clinic. Indocyanine green (Perio green, Elexxion AG, Radolfzell, Germany) prepared and applied according to manufacturer's instructions steps (mixing, application, soaking phase, rinsing, activation) in a concentration with 0.1mg/mL was administered via fine-needle syringe as the photosensitizer. Following the completion of topical application of the photosensitizer to the lesion surface, a (GaAlAs) diode laser device (Cheese Diode Laser, Wuhan Gigaa Optronics Technology Co. Ltd, China) in continuous mode (810 nm, 300 mW, 10,000 kHz, 1.26 cm2 spot area), with a 400 μm polymethylmethacrylate optical fiber tip, scanning from the periphery to the center of the lesion with an energy density of approximately 10 J/cm2 for 40 s and applied non-contact at a distance of 1 mm.
  Interventions: Combination Product: Photodynamic therapy (indocyanine green+laser)
- Control Group (No Intervention): The lesions of the patients in the control group were not treated but only followed up. Recommendations were made to reduce their pain (avoidance of hot, spicy and acidic foods, attention to oral hygiene, etc.)

INTERVENTIONS:
Combination Product: Photodynamic therapy (indocyanine green+laser) — Photodynamic therapy with indocyanine green
  Arms: Photodynamic Therapy (PDT) Group

SUMMARY:
The search for methods that can shorten the treatment process of aphthous ulcers, the etiology of which is not fully understood, continues. The aim of this study was to determine whether photodynamic therapy (PDT) is a clinically effective alternative in the treatment of oral aphthous ulcers.

DETAILED DESCRIPTION:
After sample size calculation, photodynamic therapy and control groups were formed with 15 patients with aphthous ulcer in each group. Laser therapy with indocyanine green was applied to the photodynamic therapy group on the day they were admitted to the clinic. No treatment was performed in the control group and only follow-up was performed. Lesion diameters, pain intensity and degree of improvement at the end of 1 week were recorded in all patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA-1 patients without any systemic disease,
* With a history of canker sores not exceeding 2 days,
* Not taking any antibiotics or anti-inflammatory drugs.

Exclusion Criteria:

* Laser therapy contraindicated,
* Pregnancy,
* Smoking habbit,
* Poor oral hygiene,
* Patients under 18 years of age

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Ulcer wound healing with diameter measurement | One week (preoperatively and on postoperative days 3, 5 and 7 )
  Lesion diameters were measured with a elastic ruler and the healing rate of the lesion was monitored.
Level of recovery | Postoperatively 7 th day
  A 3-point scale was used. Grade 1 represents "complete recovery", Grade 2 represents "moderate recovery", Grade 3 represents "little recovery".

SECONDARY OUTCOMES:
Pain evaluation with Visual Analogue Scale | One week
  For lesion-related pain follow-up, patients in the PDT group were asked to score the pain they felt on VAS on preoperative, 1st, 3rd, 5th and 7th days. VAS measurements of the patients in the control group were made on days 1, 3, 5 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Cennet N Eroglu, DDS,PhD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University, Van, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study published, the study information will be shared with the researchers who request it, taking into account the right to protect personal data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD and documents will be available for sharing 1 year after publication for a period of 2 years. Access to the IPD and documenta will be open on the IPDShare website with registration. The information will be freely available and can be used for any purpose. There will not be any review process or no Data Use Agreement will be necessary.
Access Criteria: IPD and documents will be available for sharing 1 year after publication for a period of 2 years. Access to the IPD and documenta will be open on the IPDShare website with registration. The information will be freely available and can be used for any purpose. There will not be any review process or no Data Use Agreement will be necessary.